CLINICAL TRIAL: NCT06767514
Title: A Randomized, Double-blinded, Multiregional Phase 3 Study of Ivonescimab Versus Pembrolizumab for the First-line Treatment of Metastatic Non-small Cell Lung Cancer in Patients Whose Tumors Demonstrate High PD-L1 Expression
Brief Title: Clinical Study of Ivonescimab for First-line Treatment of Metastatic NSCLC Patients With High PD-L1
Acronym: HARMONi-7
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMT112-3007
Record Dates: First submitted 2025-01-03; First posted 2025-01-10 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - Ivonescimab (Experimental): Subject will receive ivonescimab as an IV injection
  Interventions: Biological: Ivonescimab Injection
- Arm B - Pembrolizumab (Active Comparator): Subject will receive pembrolizumab as an IV injection
  Interventions: Biological: Pembrolizumab Injection

INTERVENTIONS:
Biological: Ivonescimab Injection — Subject will receive ivonescimab as an IV injection
  Arms: Arm A - Ivonescimab
Biological: Pembrolizumab Injection — Subject will receive Pembrolizumab as an IV injection
  Arms: Arm B - Pembrolizumab

SUMMARY:
Clinical study of ivonescimab for first-line treatment of metastatic NSCLC patients with high PD-L1. Evaluating overall survival and progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old at the time of enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 - 1
* Expected life expectancy ≥ 3 months
* Metastatic (Stage IV) NSCLC
* Histologically or cytologically confirmed squamous or non-squamous NSCLC
* Tumor demonstrates high PD-L1 expression ( TPS>50%) based on a 22C3 immunohistochemistry ( IHC) clinical assay approved / cleared by local health authorities.
* At least one measurable noncerebral lesion according to RECIST 1.1
* No prior systemic treatment for metastatic NSCLC.

Exclusion Criteria:

* Histologic or cytopathologic evidence of the presence of small cell lung carcinoma for which first-line approved therapies are indicated. For patients with non-squamous histology, actionable driver mutation testing results are required before randomization.
* Has received any prior therapy for NSCLC in the metastatic setting.
* Concurrent enrollment in another clinical study, unless patient is enrolled in a non-interventional clinical study or is completing survival follow -up.
* Known actionable genomic alterations for which first-line approved therapies are indicated
* Symptomatic CNS metastases, CNS metastasis ≥ 1.5 cm, CNS radiation within 7 days prior to randomization, potential need for CNS radiation within the first cycle, or leptomeningeal disease
* Other prior malignancy (including previously treated NSCLC) unless the patient has undergone curative therapy with no evidence of recurrence of the disease for 3 years prior to randomization
* Active autoimmune or lung disease requiring systemic therapy
* Has pre-existing peripheral neuropathy that is ≥ Grade 2 by CTCAE version 5
* Severe infection within 4 weeks prior to randomization
* Major surgical procedures or serious trauma within 4 weeks prior to randomization
* History of noninfectious pneumonia requiring systemic corticosteroids, or current interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 36 months
Progression free survival (PFS) | Up to approximately 36 months

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 36 months
Disease control rate ( DCR) | Up to approximately 36 months
Duration of response (DoR) | Up to approximately 36 months
Adverse Events (AE): incidence and severity of adverse events (AEs) and clinically significant abnormal laboratory test results | [Time Frame: From the subject signs the ICF to 30 days (AE) and 90 days (SAE related to ivonescimab/pembrolizumab ) after the last dose of study treatment or initiation of other anticancer therapy, whichever occurs first, Up to approximately 24 months.

CONTACTS AND LOCATIONS:
Locations (117):
- United States (51):
  - Clinical Study Site, Chandler, Arizona
  - Clinical Study Site, Phoenix, Arizona
  - Clinical Study Site, Hot Springs, Arkansas
  - Clinical Study Site, Cerritos, California
  - Clinical Study Site, Los Angeles, California
  - Clinical Study Site, Mountain View, California
  - Clinical Study Site, San Diego, California
  - Clinical Study Site, Aurora, Colorado
  - Clinical Study Site, Lone Tree, Colorado
  - Clinical Study Site, Loveland, Colorado
  - Clinical Study Site, Fort Lauderdale, Florida
  - Clinical Study Site, Hialeah, Florida
  - Clinical Study Site, Jacksonville, Florida
  - Clinical Study Site, Miami, Florida
  - Clinical Study Site, North Venice, Florida
  - Clinical Study Site, Orlando, Florida
  - Clinical Study Site, Pensacola, Florida
  - Clinical Study Site, Plantation, Florida
  - Clinical Study Site, Tallahassee, Florida
  - Clinical Study Site, Tamarac, Florida
  - Clinical Study Site, West Palm Beach, Florida
  - Clinical Study Site, Atlanta, Georgia
  - Clinical Study Site, Covington, Louisiana
  - Clinical Study Site, Baltimore, Maryland
  - Clinical Study Site, Boston, Massachusetts
  - Clinical Study Site, Worcester, Massachusetts
  - Clinical Study Sites, Detroit, Michigan
  - Clinical Study Site, Detroit, Michigan
  - Clinical Study Site, Saint Paul, Minnesota
  - Clinical Study Site, Kansas City, Missouri
  - Clinical Study Site, St Louis, Missouri
  - Clinical Study Site, Lebanon, New Hampshire
  - Clinical Study Site, Mullica Hill, New Jersey
  - Clinical Study Site, New Brunswick, New Jersey
  - Clinical Study Site, Glen Falls, New York
  - Clinical Study Site, Syracuse, New York
  - Clinical Study Site, Chapel Hill, North Carolina
  - Clinical Study Site, Columbus, Ohio
  - Clinical Study Sites, Lebanon, Ohio
  - Clinical Study Site, Eugene, Oregon
  - Clinical Study Site, Portland, Oregon
  - Clinical Study Site, Pittsburgh, Pennsylvania
  - Clinical Study Site, Nashville, Tennessee
  - Clinical Study Site, Austin, Texas
  - Clinical Study Site, Dallas, Texas
  - Clinical Study Site, Forth Worth, Texas
  - Clinical Study Site, Houston, Texas
  - Clinical Study Site, Tyler, Texas
  - Clinical Study Site, Webster, Texas
  - Clinical Study Site, Blacksburg, Virginia
  - Clinical Study Site, Vancouver, Washington
- Canada (3):
  - Clinical Study Site, Edmonton, Alberta
  - Clinical Study Site, London, Ontario
  - Clinical Study Site, Montreal
- China (17):
  - Clinical Study Site, Fuzhou, Fujian
  - Clinical Study Site, Guangzhou, Guangdong
  - Clinical Study Site, Haikou, Hainan
  - Clinical Study Site, Harbin, Heilongjiang
  - Clinical Site Study, Changzhou, Jiangsu
  - Clinical Study Site, Ganzhou, Jiangxi
  - Clinical Study Site, Nanchang, Jiangxi
  - Clinical Study Site, Tai’an, Shandong
  - Clinical Study Site, Weifang, Shandong
  - Clinical Study Site, Shanghai, Shanghai Municipality
  - Clinical Study Site, Kunming, Yunnan
  - Clinical Study Site, Hangzhou, Zhejiang
  - Clinical Study Site, Taizhou, Zhejiang
  - Clinical Site Study, Wenzhou, Zhejiang
  - Clinical Study Site, Changchun
  - Clinical Study Site, Guangzhou
  - Clinical Study Site, Xi'an
- France (5):
  - Clinical Study Site, Nantes, Pays de Loire
  - Clinical Study Site, Brest
  - Clinical Study Site, Créteil
  - Clinical Study Site, Marseille
  - Clinical Study Site, Paris
- Germany (3):
  - Clinical Study Site, Gauting
  - Clinical Study Site, Karlsruhe
  - Clinical Study Site, Möser
- Greece (3):
  - Clinical Study Site, Athens
  - Clinical Study Site, Rio
  - Clinical Study Site, Thessaloniki
- Clinical Study Site, Kecskemét, Hungary
- Clinical Study Site, Roma, Italy
- Clinical Study Site, Koto-Ku, Tokyo, Japan
- Mexico (4):
  - Clinical Study Site, Guadalajara
  - Clinical Study Site, Mexico City
  - Clinical Study Site, Monterrey
  - Clinical Study Site, Veracruz
- Poland (4):
  - Clinical Study Site, Lodz
  - Clinical Study Site, Lublin
  - Clinical Study Site, Poznan
  - Clinical Study Site, Skorzewo
- Romania (7):
  - Clinical Study Site, Suceagu, Cluj
  - Clinical Study Site, Baia Mare
  - Clinical Study Site, Bucharest
  - Clinical Study Site, Cluj-Napoca
  - Clinical Study Site, Craiova
  - Clinical Study Site, Iași
  - Clinical Study Site, Timișoara
- Serbia (3):
  - Clinical Study Site, Belgrade
  - Clinical Study Site, Kragujevac
  - Clinical Study Site, Novi Sad
- Spain (7):
  - Clinical Study Site, Badajoz
  - Clinical Study Site, Badalona
  - Clinical Study Site, Barcelona
  - Clinical Study Site, Girona
  - Clinical Study Site, Lugo
  - Clinical Study Site, Seville
  - Clinical Study Site, Valencia
- Turkey (Türkiye) (7):
  - Clinical Study Site, Ankara
  - Clinical Study Site, Antalya
  - Clinical Study Site, Diyarbakır
  - Clinical Study Site, Gaziantep
  - Clinical Study Site, Istanbul
  - Clinical Study Site, Konya
  - Clinical Study Site, Seyhan